CLINICAL TRIAL: NCT02447835
Title: The Effect of Short Term Atypical Antipsychotic Administration Compared to Placebo on Hepatic Insulin Extraction and Muscarinic Mediation of B-Cell Function: A Small Mechanistic, Single-Site Study
Brief Title: Effect of Short Term Atypical Antipsychotic Administration Compared to Placebo on Hepatic Insulin Extraction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Michael Rickels (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor-Investigator, Michael Rickels, Associate Professor of Medicine, University of Pennsylvania School of Medicine, Division of Endocrinology, Diabetes & Metabolism, Monell Chemical Senses Center
Organization: Monell Chemical Senses Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 815905
Record Dates: First submitted 2012-10-25; First posted 2015-05-19 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Normal Non-fluency
Keywords: Metabolic Disorders
MeSH Terms: conditions — Metabolic Diseases | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olanzapine (Active Comparator): Olanzapine administration
  Interventions: Drug: Olanzapine
- Placebo (Placebo Comparator): Placebo administration
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — Olanzapine is approved for the treatment of schizophrenia and mania associated with bipolar disorder. Olanzapine is a psychotropic agent that belongs to the thienobenzodiazepine class. The chemical designation is 2-methyl-4-4methyl-1 piperazinyl-10H-thienol (2,3-b)[1,5]benzodiazepine. The molecular formula is C17H20N4S which corresponds to a molecular weight of 312.44.Olanzpine is a yellow crystalline solid which is practically insoluble in water. Olanzapine is a selective monoaminergic antagonist with high affinity binding to the following receptors:5HT2A2C, 5HT6, dopamine 2-4, histamine H1, and adrenergic α-1. In addition olanzapine is an antagonist with moderate affinity for muscarinic M1-5 and 5HT3. The mechanism of action of olanzapine is unknown although it may be mediated through a combination of dopamine and serotonergic type 2 receptors.
  Other Names: Zyprexa

SUMMARY:
Within the past 20 years, there has been a striking increase in the incidence of obesity 1;2, type 2 diabetes mellitus (T2DM) 3-5, and cardiovascular diseases (CVD) in the schizophrenic population 6-8 . Large NIH-funded trials indicate that the prevalence of metabolic syndrome is twice to three times greater in schizophrenic patients on a specific class of drug termed the "atypical antipsychotics" (AAPs), of which olanzapine is an example, as compared to matched controls 8. Identification of the pathophysiological mechanisms contributing to metabolic disease in schizophrenic patients on AAPs has been hampered by the inability to differentiate underlying disease from treatment-emergent complications. In addition, despite falling within the same drug class, different AAPs exhibit differential associations with metabolic disease. Olanzapine is one of the AAPs associated with the greatest weight gain and degree of metabolic impairments.

DETAILED DESCRIPTION:
The increased incidence of T2DM and CVD with the AAPs has been assumed a consequence of weight gain. However, accumulating evidence of weight-independent effects derived from in vitro and rodent studies suggests a direct effect of some AAPs on the pancreatic B-cell and the liver. We have recently completed the first of two studies supported by an NIH grant which provides evidence for a direct effect of olanzapine on metabolism, independent of weight gain or psychiatric disease. Findings from the first study indicate that short-term administration (9-days) of olanzapine compared to aripiprazole, another AAP as well as placebo dramatically increases post-prandial insulin levels in healthy control subjects independent of weight gain; providing evidence of tissue specific effects of the drug in humans. We also found that the increase in insulin was not accompanied by an increase in plasma C-peptide concentrations suggesting that olanzapine may decrease hepatic insulin extraction. Decreases in hepatic insulin extraction can be mediated through muscarinic blockade and in fact, data from our laboratory demonstrates that atropine (the muscarinic antagonist) inhibits hepatic insulin extraction in humans. Blockade of muscarinic receptors is consistent with the receptor binding profile of olanzapine which shows a higher receptor antagonism for muscarinic receptors compared to other AAPs. In addition, we also found significant increases in glucagon-like peptide 1 (GLP-1) and decreases in insulin sensitivity following olanzapine administration compared to aripiprazole and placebo. The proposed study follows up on these findings with a study designed to investigate the mechanisms contributing to the olanzapine-induced post-prandial hyperinsulinemia and GLP-1. The overall hypothesis of this study is that olanzapine blocks peripheral muscarinic receptors, leading to a compensatory increase in vagal efferent activation which contributes to an increase in insulin secretion.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ages 18-40
2. BMI 19-24.5kg/m2
3. Systolic BP <130mm Hg
4. Diastolic BP <85mm Hg
5. Subjects capable of giving informed consent, with no past or present psychiatric history
6. Only women on oral contraceptives with constant dosing regimens or Depo-Provera for >3 months, to ensure uniform hormonal delivery throughout the study duration
7. No medications except as above noted
8. Weight stable
9. Minimal exercise regime that includes walking, running or biking

Exclusion Criteria:

1. History of heart disease, colitis, autonomic neuropathy, hepatic or renal disease
2. DSM-IV diagnosis of past or present psychiatric history, including clinically significant depression
3. Drug/Alcohol dependence, homelessness, or inability to give informed consent
4. History of asthma, congenital obstructive bladder, peptic ulcer, vasomotor instability, epilepsy, Parkinsonism, elevated thyroid hormone levels
5. Diagnosis of diabetes
6. BMI>25 kg/m2
7. Prescription medication (excluding the contraceptive methods described above)
8. Hemoglobin <11
9. Abnormal laboratory tests which are clinically significant per the investigator
10. Females pregnant or lactating
11. Females: not taking hormonal contraceptives; taking hormonal contraceptives of varying dosage throughout the month
12. Currently on a weight loss diet
13. Moderate to significant exercise regime that includes swimming, weight lifting or other form of exercise not reproducible within CTRC.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Determine the vagal contribution to the olanzapine-induced increase in circulating insulin levels. | 12 days

SECONDARY OUTCOMES:
Determine if olanzapine increases meal-related/satiety peptides | 12 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States